CLINICAL TRIAL: NCT00388986
Title: An Open-label, Crossover Study to Investigate the Potential Pharmacodynamic and Potential Pharmacokinetic Interaction Between Glyburide and GK Activator(2) in Type 2 Diabetes Patients Inadequately Controlled With Glyburide as Standard Prescribed Therapy.
Brief Title: A Drug-Drug Interaction Study of GK Activator (2) and Glyburide in Patients With Type 2 Diabetes.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NP20194
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glyburide

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: GK Activator (2); Drug: Glyburide
- 2 (Experimental)
  Interventions: Drug: GK Activator (2)
- 3 (Experimental)
  Interventions: Drug: Glyburide

INTERVENTIONS:
Drug: GK Activator (2) — 100mg po bid
  Arms: 1; 2
Drug: Glyburide — 10-20mg po daily
  Arms: 1; 3

SUMMARY:
This study will assess the potential pharmacodynamic and potential pharmacokinetic interaction between GK Activator (2) and glyburide, in type 2 diabetes patients not adequately controlled with glyburide as standard prescribed therapy. Patients will enter the study taking a dose of glyburide (10-20mg po daily) as prescribed prior to study start. GK Activator (2) 100mg bid will be added for 5 days. From days 6-12 patients will receive GK Activator (2) monotherapy, and from day 13 GK Activator (2) will be discontinued and glyburide treatment re-started. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, aged 18-75 years;
* type 2 diabetes mellitus; currently on glyburide 10-20 mg/day for >=3 months;
* untreated, or taken off anti-diabetic or statin therapy >=2 weeks before study start.

Exclusion Criteria:

* type 1 diabetes mellitus, or latent autoimmune diabetes in adults;
* diabetic neuropathy, retinopathy or nephropathy;
* patients treated with insulin or PPAR gamma agonist with 6 weeks of screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
AUC0-6h of plasma glucose | Days -1, 6 and 12
AUC0-12h of GK Activator (2) and metabolite. | Days 6 and 12
AUC0-tau of glyburide | Days -1 and 6

SECONDARY OUTCOMES:
AEs, laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United States (4):
  - Cypress, California
  - Honolulu, Hawaii
  - Buffalo, New York
  - San Antonio, Texas